CLINICAL TRIAL: NCT05892159
Title: Heart Rate Variability Biofeedback in the Treatment of Ulcerative Colitis
Brief Title: Heart Rate Variability (HRV) Biofeedback to Treat Ulcerative Colitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Robert Hirten, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-21-00870
Record Dates: First submitted 2023-05-28; First posted 2023-06-07 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRV biofeedback (Experimental): An HRV biofeedback tool will be employed in which individuals will breathe at their resonance frequency to optimize HRV and autonomic nervous system signatures.
  Interventions: Behavioral: HRV biofeedback

INTERVENTIONS:
Behavioral: HRV biofeedback — An HRV biofeedback tool will be employed and utilized by individuals each day for the first 5 weeks during the intervention period.

SUMMARY:
This is a prospective interventional study exploring the modifiability of physiological metrics, namely Heart Rate Variability (HRV), using a 5-week standardized HRV biofeedback intervention in subjects with symptomatic ulcerative colitis. Participants will be followed for 17 weeks. The goal is the understand if modifying these markers can impact ulcerative colitis related symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (18-65 years old)
* Ulcerative colitis with a symptomatic flare (SCCAI ≥3) and without inflammation (FC<250µg/ml)

Exclusion Criteria:

* Individuals who take medications known to alter heart rate variability
* Individuals with pacemakers or other implantable devices

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-02-27 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
Irritable Bowel Syndrome Symptom Severity Scale Score | at end of Week 5
  Clinical symptom improvement: Improvement in a clinical symptom score. Responders will be classified as those with an Irritable Bowel Syndrome Symptom Severity Scale (IBS-SSS; full scale range 0-500, where severe symptoms are ≥ 300) that decreases by ≥ 50 points at the end of week 5.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hirten, Principal Investigator — Icahn School of Medicine at Mount Sinai

IPD SHARING:
Plan to Share IPD: No
There are limitations in our institutional review board approval relating to individual patient level data sharing.